CLINICAL TRIAL: NCT02527928
Title: Cost-Effectiveness of Different Formulation of Amphotericin B in Private and Public Hospitals in Southern Brazil
Brief Title: Cost-Effectiveness of Amphotericin B
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospital Universitario Evangelico de Curitiba (Other)
Responsible Party: Principal Investigator, Felipe Francisco Bondan Tuon, MD, Hospital Universitario Evangelico de Curitiba
Other Study IDs: teva
Record Dates: First submitted 2015-03-20; First posted 2015-08-19 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Invasive Fungal Infections
Keywords: pharmacoeconomics
MeSH Terms: conditions — Invasive Fungal Infections

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- desoxycholate: Amphotericin B desoxicholate
  Interventions: Other: None intervention
- Anfolipidcomplex: Amphotericin B complex lipid
- ABLiposomal: Amphotericin B liposomal

INTERVENTIONS:
Other: None intervention
  Groups: desoxycholate

SUMMARY:
Invasive fungal infections (IFIs) are complications that happen in the hospital, usually in patients hospitalized for long periods in intensive care units (ICU) after invasive procedures, and in specific populations, such as cancer patients. The aim of this study is to determine the direct and indirect hospital costs with different formulations of amphotericin B (deoxycholate, lipid complex and liposomal) in different public and private hospitals in the city of Curitiba, Paraná, Brazil.

DETAILED DESCRIPTION:
BACKGROUND There are several American studies on the costs that the antifungal represents in the hospital bills, but in Brazil we do not have this type of study (WINGARD 2007; GREENE 2007). The American studies cannot be extrapolated to Brazil because the cost of drugs is different as well as other hospital charges. Furthermore, in Brazil spending on public medicine, governed by the Unified Health System (SUS) are different from those employed in the complementary health services (private health services). For these reasons, knowledge of the percentage they represent in the antifungal hospital bills in order to define the actual cost-effectiveness of different formulations of amphotericin B, considering length of hospital adverse events and mortality is needed.

OBJECTIVES:

Determine the direct and indirect hospital costs with different formulations of amphotericin B (deoxycholate, lipid complex and liposomal) in different public and private hospitals in the city of Curitiba, Paraná, Brazil.

Specifics

1. Measuring the total cost of hospitalization with antifungal treatment.
2. Measure the direct spending each formulation of amphotericin B
3. Measuring the indirect costs related to the nephrotoxicity of different formulations of amphotericin B
4. Assemble a model of cost-effectiveness of different formulations of amphotericin B

METHODS

This is a retrospective, observational, cohort study economic. Database of admissions of patients who used antifungal in all private hospital from an specific private health system (more than 5 hospitals) and databases of two large public hospitals in Curitiba (Evangelical University and the Clinical Hospital).

Patients over 18 years of age who used any formulation of amphotericin B will be included.

The data will be evaluated by the principal diagnosis ICD10 obtained at admission or discharge, the total length of stay, length of hospital stay before antifungal start, length of stay after initiation of antifungal drug, which formulation of amphotericin B used, the necessity and amount of dialysis. Also we will assess the final outcome of the patient (death or cure). Other epidemiological data such as age and gender will be evaluated.

A cost analysis will be based on total bill of the patient, the cost of antifungal, cost throughout the dialysis procedure, cost of laboratory tests used in monitoring during treatment with amphotericin (complete blood count, electrolytes, renal function, partial urine, function liver, electrocardiogram). The cost will be measured in American Dollar. These data were obtained from a similar study used for costing with antifungals in invasive aspergillosis in the USA (KIM 2011).

Data will be analyzed according to the type of variable. Means or medians will be used for continuous variables with standard deviation. Statistical methods for comparing means or medians will be parametric or non-parametric, as well as chi-square test for dichotomous variables. The data will be considered statistically significant when a difference of 5% (p <0.05) occur. Other multivariable method can be applied according with the results.

Informed consent is not necessary because is a retrospective cohort with data obtained from medical charts, without any intervention.

Principal investigator and co-investigator will be the sponsor for fill the request. All the survey will be fulfilled by investigator and co-investigator. The survey is attached in the end of the project.

This study will be sent for ethics committee for approval before start.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age who used any formulation of amphotericin B will be included

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a study of pharmacoeconomics. Patients who used amphotericin B e total cost of hospitalization.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-09; Primary Completion 2015-12 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Cost | Fungal infection at day 100
  The outcome will measured in US dollar.